CLINICAL TRIAL: NCT03427892
Title: Brexpiprazole for Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102016-048
Record Dates: First submitted 2016-12-28; First posted 2018-02-09 (Actual); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Bipolar Depression
Keywords: mood; bipolar; depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brexpiprazole (Experimental): Brexipiprazole will be taken orally beginning at 0.5 mg/day with an increase to 1 mg/day at week 1 and 2 mg/day at week 2. If reduction in mood symptoms does not occur, the dose will increase to 3 mg/day and 4 mg/day.
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Brexpiprazole is an atypical antipsychotic drug that is used to treat mental/mood disorders.
  Other Names: Rexulti

SUMMARY:
The investigators will conduct an 8-week, non-randomized, open-label study of brexpiprazole in 20 persons with bipolar I or II disorder, depressed mood state. Primary aim will be to assess if brexpiprazole is associated with a reduction in depressive symptom severity using the Montgomery-Asberg Depression Rating Scale (MADRS). Secondary aims will include an assessment of the following in patients with bipolar disorder taking brexpiprazole: manic symptoms, cognition, safety and tolerability of brexpiprazole, and quality of life.

Subjects will be discontinued from the study if any of the following conditions occurs: change in diagnosis to other than bipolar I or II disorder, development of active suicidal or homicidal ideation with plan and intent, worsening of mood symptoms, that in the opinion of the investigators requires discontinuation, pregnancy, development of severe life-threatening medical condition, involuntary psychiatric hospitalization or incarceration.

DETAILED DESCRIPTION:
We will conduct an 8-week, non-randomized, open label study of brexpiprazole in 20 persons with bipolar disorder. Primary Aim will be to determine if brexpiprazole is associated with a reduction in depressive symptom severity using the Montgomery-Asberg Depression Rating Scale (MADRS) in outpatients with bipolar disorder, depressed mood state. Secondary Aims will be: 1) Assess manic symptoms in patients with bipolar disorder receiving brexpiprazole, 2) Assess cognition in patients with bipolar disorder receiving brexpiprazole, 3) Assess the safety and tolerability of brexpiprazole in patients with bipolar disorder, 4) Assess quality of life in patients with bipolar disorder receiving brexpiprazole. Subjects will be discontinued from the study if any of the following conditions occurs: change in diagnosis to other than bipolar I or II disorder, development of active suicidal or homicidal ideation with plan and intent, worsening in mood symptoms, that in the opinion of the investigators requires discontinuation, pregnancy, development of severe or life-threatening medical condition, involuntary psychiatric hospitalization or incarceration.

Study Procedures:

Baseline: This visit will be split into two portions: Baseline 1 and Baseline 2.

For Baseline 1 (~3 hours), the psychiatric diagnosis will be confirmed by the structured clinical interview for DSM-5 (SCID), mood assessed via the Montgomery-Asberg Depression Rating Scale (MADRS), depression via the Inventory of Depressive Symptomatology Self-Report (IDS-SR30), mania via the Young Mania Rating Scale, and quality of life via the Quality of Life in Bipolar Disorder (QOLBD). Blood will be drawn for complete blood count (CBC), Comprehensive Metabolic Panel (CMP, includes a liver panel with AST, ALT, as well as lipids), and high-sensitivity c-reactive protein (hs-CRP). A urine sample for drug screen and pregnancy test (if applicable), psychiatrist assessment, physical exam, collection of weight and vitals will be completed.

For Baseline 2 (~2 hours), recent depressive symptoms will be assessed via the IDS-SR30 and MADRS, mania via the YMRS, current mood via Internal State Scale (ISS), suicidal ideation will be assessed via the Columbia Suicide Severity Rating Scale (CSSRS), safety and side effects will be assessed with the SAFTEE, the Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Scale (BAS) and Simpson-Angus Scale (SAS). Subjects will also complete the The Ray Auditory Verbal Learning Test (RAVLT) to assess word memory, the Stroop test to measure attention, speed, and accuracy of thinking, and The Trail Making Test (TMT) to measure attention, speed and accuracy. A urine sample for drug screen and pregnancy test (if applicable) will also be completed. Brexpiprazole capsules will be initiated at 0.5 mg/day.

Baseline 2 to Week 1: Subjects will be given the ISS to fill out at home. Subjects will be asked to complete the scale at home on 7 consecutive days between Baseline 2 and Week 1 visits and return the filled out scales to the researcher's office. The scale will take approximately 3-5 minutes to fill out.

Week 1, 2, 3, 6 (~1.5 hours each): Subjects will complete the MADRS, YMRS, IDS-SR30, ISS, SAFTEE, CSSRS, AIMS, BAS, SAS, and a urine sample will be collected for a drug screen. Subjects will meet with the psychiatrist for weekly assessment and vitals will be collected.

Week 4 (~2 hours): Subjects will complete the MADRS, IDS-SR, YMRS, SAFTEE, ISS, C-SSRS, AIMS, BAS, SAS, RAVLT, Stroop, TMT, vital signs, a urine sample for a drug screen and a urine pregnancy test, and visit the doctor for a psychiatric evaluation.

Week 8 (final visit ~2.5 hours): Subjects will complete the MADRS, IDS-SR, YMRS, SAFTEE, ISS, C-SSRS, AIMS, BAS, SAS, RAVLT, Stroop, TMT, QOLBD, vital signs, a urine sample for drug screen, take a urine pregnancy test, have blood drawn for clinical testing (CBC, CMP, hs-CRP), and visit the doctor for a psychiatric evaluation and physical exam. During this visit, participants will also be provided with aftercare referral information and will begin their medication taper. The medication taper schedule is described below under "Study Medication and Intervention Description".

Safety Phone Call (~15 min): Participants will receive a phone call from researchers 7-10 days following their Week 8 study visit (at the end of their tapering schedule). During this phone call, the researchers will assess any withdrawal effects or adverse events and check on the status of the aftercare referrals.

Participants will be paid for their time and inconvenience per visit as follows: $60 at Baseline 1, Baseline 2, weeks 1, 2, 3, 6; $70 at week 4; $90 for week 8. Participants will also be paid for each ISS scale they bring back at the rate of $1 per scale (maximum $7). These payments will be processed during Week 1 visit. These payments will be completed via the ClinCard system. Bus or rail passes will be provided. After study completion, standard psychiatric care will be provided until referral is arranged.

Study Medication and Intervention Description:

Participants will be initiated on a 0.5 mg/day brexpiprazole dose (week 0/baseline); after one week the dose will be increased to 1 mg/day (week 1), after another week to 2 mg/day (week 2). If any dose appears to be poorly tolerated, the dose titration can be slowed or stopped based on clinician judgment. If response in weeks 3-6, defined as a 50% reduction in the MADRS, has not been achieved, and the current dose is well tolerated, then additional dose increases to 3 mg/day and 4 mg/day (maximum allowed dose in protocol) will occur with at least a one week interval between dose increases.

Following the last study visit (Week 8), participants will be gradually tapered off the medication every 2 days until they stop taking the medication completely. For example, if a participants takes 4 mg of brexpiparzole at Week 8, then he/she will take 3 mg for 2 days, then 2 mg for 2 days, then 1 mg for 2 days, and then 0.5 mg for 2 days. At the end of the tapering period (7-10 days depending on the highest brexpiprazole dose at the end of the study), participants will receive a safety phone call from a research staff member to assess any withdrawal symptoms and check on the status of the aftercare referrals.

Biostatistics:

Primary Aim: Determine if brexpiprazole is associated with a reduction in depressive symptom severity in outpatients with bipolar disorder, depressed mood state.

1. The MADRS will be the primary outcome measure with the IDS-SR as a secondary outcome measure. Weekly scores on the MADRS and IDS-SR will be assessed using one-way repeated measures. Analysis of Covariance (rm-ANCOVA), controlling for age and sex as potential confounding variables, with time as the main effect. Participants will be included if they complete one post-baseline assessment (intent-to-treat sample). In addition, rates of depression response (≥ 50% reduction from baseline) and remission (≤10 on the MADRS and ≤12 on the IDS-SR) will be assessed. A significance level of 0.05 will be set for all analyses, with all tests being two-tailed.

   Secondary Aims:
2. Assess manic symptoms in patients with bipolar disorder receiving brexpiprazole. YMRS scores will be assessed as with the primary aim above.
3. Assess cognition in patients with bipolar disorder receiving brexpiprazole. Scores on the RAVLT, Stroop and TMT will be assessed at baseline compared to weeks 4 and 8 separately using paired t-tests or paired-sample Wilcoxon Signed Rank test.
4. Assess the safety and tolerability of brexpiprazole in patients with bipolar disorder. Scores on the SAFTEE, C-SSRS, AIMS, BAS and SAS will be assessed as with the primary aim.
5. Assess quality of life in patients with bipolar disorder receiving brexpiprazole. The QOLBD will be assessed as above for cognition.
6. Assess peripheral inflammation in patients with bipolar disorder receiving brexpiprazole. Values on hs-CRP will be compared between baseline and exit as with cognition above.
7. Assess relationships between changes in outcomes measures. Correlations between outcome measures (e.g. depressive symptoms and cognition, depressive symptoms and inflammation) will be assessed using Pearson's or Spearman's correlation coefficients.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient men and women ages 18-65
* Bipolar I or II disorders, currently depressed mood state based on a SCID for DSM-5; Mixed features in DSM-5 are allowed, but those with a Young Mania Rating Scale score ≥ 15 will be excluded
* Baseline MADRS score ≥ 20

Exclusion Criteria:

* Mood disorders other than bipolar I or II disorders (e.g., bipolar NOS, or cyclothymic disorders, schizophrenia, schizoaffective disorder, or unipolar depression based on the SCID), other disorders, e.g. anxiety disorders, will be allowed
* Current (last 14 days) treatment with an antipsychotic or antidepressant
* History of neuroleptic malignant syndrome or tardive dyskinesia
* Prior history of brexpiprazole use
* Vulnerable populations (e.g., pregnant, nursing, cognitively impaired, incarcerated)
* High risk for suicide defined as > 1 attempt in past 12 months that required medical attention, any attempt in the past 3 months or current suicidal ideation with plan and intent such that outpatient care is precluded
* Severe or life-threatening medical condition, or laboratory or physical examination findings consistent with serious medical illness (e.g., dangerously abnormal electrolytes)
* Moderate or severe hepatic or renal impairment based on medical history and laboratory analyses
* Taking moderate or strong induces or inhibitors of CYP2D6 or CYP3A4

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, M.D., Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scala M, Biondi L, Fabbri C, Serretti A. Efficacy of Brexpiprazole Combination Therapy on Anhedonia in a Case of Treatment Resistant Bipolar II Depression. J Clin Psychopharmacol. 2023 Sep-Oct 01;43(5):453-455. doi: 10.1097/JCP.0000000000001732. Epub 2023 Jul 14. No abstract available. PMID 37683234

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients recruited through flyers and other forms of advertisement. Patients met DSM-5 criteria for bipolar I or II disorder, with a current moderate to severe depressed mood state. The last patient completed on March 15, 2018.
Pre-assignment Details: Of the 30 patients consented and screened during the duration of the study between March 2017 and December 2017, 9 screen failed and 21 were enrolled within the study. The study was non-randomized and all patients received the same study condition.
Period: Overall Study
Arm/Group | Brexpiprazole
Started (Open Label (baseline to week 8)) | 21
Completed | 19 (Of the 21 recruited, 19 completed at least one post baseline visit, included in the analysis.)
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.74 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 9
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19
Montgomery Asberg Depression Rating Scale (MADRS) score ranges from 0-60, higher score is indicative [Mean (Standard Deviation); unit: units on a scale] — Montgomery Asberg Depression Rating Scale (MADRS) score ranges from 0-60, higher score is indicative of more acute depressive symptoms."
  units on a scale | 31.95 (10.33)

OUTCOME MEASURES:

1. Primary Outcome: The Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The Montgomery-Asberg Depression Rating Scale is used to assess depressive symptom severity. There are 10 items and each item is rated from 0 to 6 (increasing severity) based on the assessment of symptoms within the past 7 days. Scoring is assisted by descriptive anchors that serve as useful guides at 0,2,4, 8. Odd numbers (1,3,5) between the descriptive anchors are also meant to be scored. Highest possible MADRS score is 60. Lowest possible MADRS score is 0. MADRS is scored by taking the sum of the scores for each item. A higher score is indicative of more acute depressive symptoms.
Time Frame: Baseline through week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 19
score on a scale
  MADRS Baseline | 31.95 (10.33)
  MADRS Week 4 | 9.95 (8.28)
  MADRS Week 8 | 10.95 (9.59)
Statistical Analysis 1: Comparison: Brexpiprazole; Primary Aim is to determine if brexpiprazole is associated with a reduction in depressive symptom severity in bipolar disorder outpatients. A sample size of 17 provides 80% power for a paired t-test to compare baseline to exit change scores on the MADRS of 7 (SD 10) (a more conservative change than with even the low 1 mg dose of brexpiprazole in Thase et. al. (2015)) with alpha=.05. A sample size of n=20 will allow for some early withdrawals without postbaseline data (10); Test type: Other — Within subjects design; single group. Intent-to-treat (ITT) sample was used in the analysis, such that all participants who completed the baseline visit and at least one post-baseline assessment were included in the analysis; p < .001, ANOVA — To analyze mood symptoms, cognitive performance, and side effects, separate one-way repeated measures analyses of variance (ANVOA) were performed. Time (bsl, wk 4, and wk 8) was included as the within-subject factor; One-way repeated measures analyses of variance (ANVOA) were performed. Time (bsl, wk 4, wk8) was included as the within-subject factor

2. Secondary Outcome: Young Mania Rating Scale (YMRS)
Description: Young Mania Rating Scale is an observer-rated measure of mania symptoms. It has 11 items and each items has 5 defined anchor points with increasing severity that describe the symptom characteristics. YMRS is scored by taking sum of the scores for the 11 items. A higher score indicative of more acute manic symptoms. Seven of the items are scored between 0 and 4. Four items allow for scoring between anchor points (ranging 1 to 8). Maximum score is 60 and minimum score is 0.
Time Frame: Baseline through week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 19
score on a scale
  YMRS Baseline | 4.63 (3.22)
  YMRS Week 4 | 4.21 (3.97)
  YMRS Week 8 | 4.42 (5.36)
Statistical Analysis 1: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .93, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Rey Auditoy Verbal Learning Test
Description: Rey Auditory Verbal Learning Test (RAVLT) is a test of verbal learning and declarative memory. During the test, 15 nouns that are read aloud for 5 consecutive trials. Each trial is followed by a free recall test (participant is asked to recall the words that were just read to them). The sum of correctly recalled words across 5 trials is called the total raw score. On completion of Trial 5, an interference list of 15 words (List B) is presented, followed by a free recall test of that list. After a 20-min delay, the examinee is again required to recall the words from list A - this is called the delay raw score. The raw scores on both the total recall and the delay trials (number of words correct across trials 1-5) are converted to standardized T-scores (Mean=50; SD=10; range 20-100) based on participant age and gender. The scores below are presented as T-scores, with higher scores indicative of better performance.
Time Frame: Baseline through week 8
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 19
T-scores
  RAVLT T Score Baseline | 37.47 (16.67)
  RAVLT T Score Week 4 | 37.79 (10.36)
  RAVLT T Score Week 8 | 40.42 (11.97)
  RAVLT Delay Baseline | 39.74 (13.23)
  RAVLT Delay Week 4 | 37.00 (9.010)
  RAVLT Delay Week 8 | 39.26 (13.14)
Statistical Analysis 1: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .49, ANOVA — To analyze mood symptoms, cognitive performance, and side effects, separate one-way repeated measures analyses of variance (ANVOA) were performed. Time (bsl, wk 4, and wk 8) was included as the within-subject factor. The above reported is RAVLT Score; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .56, ANOVA — Within subjects design; single group. Intent-to-treat (ITT) sample was used in the analysis, such that all participants who completed the baseline visit and at least one post-baseline assessment were included in the analysis.Reported is delay score; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Stroop Task
Description: The Stroop task evaluates attention, speed, and accuracy of thinking. Stroop task consists of three separate trials: word, color, and color-word (CW) naming. For each trial, a raw score (correct number of words named) is recorded. The raw score for each trial is converted to a T-score based on participant's age and education level. The possible T-scores range from 15-85 for the word trial, 8-92 for the color trial, and 3-98 for the color-word trial. The interference score (Inter) is also derived from the color-word score, with T-scores ranging from 21-80. Higher numbers indicate better performance. The entered values represent T-scores.
Time Frame: Baseline through week 8
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 19
T-scores
  STROOP-CW Baseline | 48.11 (7.39)
  STROOP-CW Week 4 | 41.21 (34.73)
  STROOP-CW Week 8 | 50.74 (6.82)
  STROOP-Inter Baseline | 49.89 (5.64)
  STROOP-Inter Week 4 | 43.47 (34.95)
  STROOP-Inter Week 8 | 51.79 (5.06)
Statistical Analysis 1: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .221, ANOVA — To analyze mood symptoms, cognitive performance, and side effects, separate one-way repeated measures analyses of variance (ANVOA) were performed. Time (bsl, wk 4, and wk 8) was included as the within-subject factor. Reported is CW score; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .306, ANOVA — To analyze mood symptoms, cognitive performance, and side effects, separate one-way repeated measures analyses of variance (ANVOA) were performed. Time (bsl, wk 4, and wk 8) was included as the within-subject factor.Reported is Inter. score; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Trail Making Test (TMT)
Description: The Trail Making Test (TMT) measures attention, speed, and accuracy. TMT consists of two parts: Trails A and Trails B. The performance on each test is measured in seconds and represents how quickly a participant can connect the numbers (Trails A) and the numbers and letters (Trails B) together. The number of seconds it takes to complete each part of TMT is converted to a T-score based on gender, age, race, and education. The T-scores range from 0-100 with higher scores indicating better (faster) performance. The entered data are presented as T-Scores.
Time Frame: Baseline through week 8
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 19
T-scores
  TMT A Score Baseline | 47.74 (9.34)
  TMT A Score Week 4 | 51.16 (11.49)
  TMT A Score Week 8 | 53.47 (13.24)
  TMT B Score Baseline | 45.79 (6.39)
  TMT B Score Week 4 | 47.37 (7.57)
  TMT B Score Week 8 | 49.68 (11.48)
Statistical Analysis 1: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .07, ANOVA — To analyze mood symptoms, cognitive performance, and side effects, separate one-way repeated measures analyses of variance (ANVOA) were performed. Time (bsl, wk 4, and wk 8) was included as the within-subject factor. The above reported is TMT A; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .19, ANOVA — To analyze mood symptoms, cognitive performance, and side effects, separate one-way repeated measures analyses of variance (ANVOA) were performed. Time (bsl, wk 4, and wk 8) was included as the within-subject factor.The above reported is TMT B; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Systematic Assessment For Treatment Emergent Events
Description: The Systematic Assessment for Treatment Emergent Effects (SAFTEE) is a self-report scale used in clinical trials and is designed to evaluate the degree to which each possible side effect is bothersome to a participant. There are 55 items on the scale (each item represents a different side effect), with each item rated on a 4-point scale such as "not bothersome - 0 (zero)", "mildly bothersome - 1", "moderately bothersome - 2", "severely bothersome - 3". The total possible range of scores on the scale is 0-165. The higher scores indicate a higher degree of being bothered by various side effects.
Time Frame: Baseline through week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 19
score on a scale
  SAFTEE Baseline | 49.79 (27.74)
  SAFTEE Week 4 | 23.53 (20.51)
  SAFTEE Week 8 | 23.42 (22.24)
Statistical Analysis 1: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < .001, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Columbia Suicide Severity Rating Scale
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) is a structured interview and rating scale used to measure suicidal thoughts and behaviors. Actual attempts, interrupted attempts, and aborted attempts are measured as positive integers (zero and above). The minimum value for the actual, interrupted, and aborted attempt is zero (reflecting no past suicidal behavior). There is no maximum scale value, as the number of attempts differs for each participant. The entered values represent the average number of actual, interrupted, and aborted attempts in the group. Higher values reflect a higher number of attempts experienced by each participant (equivalent to a worse outcome).
Time Frame: Baseline through week 8
Measure: Mean (Standard Deviation); unit: attempts
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 19
attempts
  C-SSRS Actual Attempts -in lifetime- Baseline | 1.35 (2.43)
  C-SSRS Actual Attempts-since last visit Week 4 | 0.00 (0.00)
  C-SSRS Actual Attempts-since last visit Week 8 | 0.00 (0.00)
  C-SSRS Interrupted Attempts-in lifetime- Baseline | 0.10 (0.31)
  CSSRS Interrupted Attempts-since last visit Week 4 | 0.00 (0.00)
  CSSRS Interrupted Attempts-since last visit Week 8 | 0.00 (0.00)
  C-SSRS Aborted Attempt-in lifetime-Baseline | 0.00 (0.00)
  C-SSRS Aborted Attempt-since last visit-Week 4 | 0.00 (0.00)
  C-SSRS Aborted Attempt-since last visit-Week 8 | 0.00 (0.00)
Statistical Analysis 1: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .022, ANOVA — To analyze separate one-way repeated measures analyses of variance (ANOVA) were performed. Time (baseline, week 4, week 8) was included as the within-subject factor.Above is from baseline to week 8 for C-SSRS AA, IA, and ABA; One-way repeated measures (ANOVA) were performed. Time (baseline, wk 4, wk 8) included as within-subject factor. Above is for C-SSRS AA,IA, and ABA
Statistical Analysis 2: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .163, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

8. Secondary Outcome: Abnormal Involuntary Movement Scale
Description: The Abnormal Involuntary Movement Scale (AIMS) is an assessment of movements to determine any long-term drug induced movement disorders.There are 10 items on the scale with scores ranging from 0-4 (0 None/Normal, 1 minimal, 2 mild, 3 moderate,4 severe). 4 items assess facial and oral movements, 2 items measure extremity movements, 1 item measures trunk movements, and 3 items measure global judgments regarding symptoms assessed. A total score is the sum of scores for items assessing facial and oral movements, extremity movements, and trunk movement (scores ranging from 0-28), with 0 being the lowest score, and 28 being the highest score. A higher score is indicative of a higher severity in symptomatology.
Time Frame: Baseline through week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 19
score on a scale
  AIMS Baseline | 0.63 (2.09)
  AIMS Week 4 | 1.26 (2.23)
  AIMS Week 8 | 1.16 (2.29)
Statistical Analysis 1: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .133, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

9. Secondary Outcome: Barnes Akathisia Scale
Description: The Barnes Akathisia Scale (BAS) is an assessment of movements to determine any short-term drug-induced movement disorders. There are 5 items.Items 1-3 are rated from a scale of 0-3 with 0 indicating the least severity, and 3 indicating the highest severity of symptoms. Item 4 is a global assessment of symptoms assessed and the severity is assessed on a scale of 0-5, with 0 indication least severity and 5 indicating the most severity.The total score is the sum of all the item scores (scores ranging from 0-14).With higher scores reflecting worse outcome.
Time Frame: Baseline through week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 19
score on a scale
  BAS Baseline | 0.12 (0.12)
  BAS Week 4 | 2.37 (0.56)
  BAS Week 8 | 2.47 (0.57)
Statistical Analysis 1: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .002, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

10. Secondary Outcome: Simpson Angus Scale
Description: The Simpson Angus Scale (SAS) measured drug-induced movement side effects. There are 10 items on the scale, with each item scored on a scale of 0-4 (least to most severe). The total possible range of scores across all items is 0-40, with higher scores indicative of worse outcome.
Time Frame: Baseline through week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 19
score on a scale
  SAS Baseline | 0.37 (0.23)
  SAS Week 4 | 1.16 (0.34)
  SAS Week 8 | 1.00 (0.32)
Statistical Analysis 1: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .002, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

11. Secondary Outcome: Quality of Life in Bipolar Disorder (QOLBD)
Description: The Quality Of Life in Bipolar Disorder (QOLBD) is a measure of the quality of life in patients with bipolar disorder. All questions on the scale ask about a range of experiences, behaviors, and feeling related to the quality of life. For each question, a participant is asked to indicate how much they agree with each question. The scale consists of 12 questions, with each question measured on a 5-point scale, such as "strongly disagree - 1", "disagree - 2", "neutral - 3", "agree - 4", "strongly agree - 5". The total possible range of scores on the scale is 12-60. Higher scores indicate better quality of life.
Time Frame: Baseline and at week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 19
score on a scale
  QOLBD baseline | 30.38 (8.97)
  QOLBD Week 8 | 40.95 (11.03)
Statistical Analysis 1: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .005, t-test, 2 sided — Pairwise comparisons were also performed to determine which time points were significantly different from one another. Baseline to week 8 is reported above; Pairwise comparisons were also performed to determine which time points were significantly different from one another

12. Secondary Outcome: The Inventory of Depressive Symptomatology Self-Report (IDS-SR30)
Description: An 30 item inventory self report assessing depressive symptoms and mood, within the past seven days. With the score range of 0-90 with higher scores indicating worse outcome.
Time Frame: Baseline through week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 19
score on a scale
  IDS-SR30 Baseline | 41.63 (17.50)
  IDS-SR30 Week 4 | 18.95 (12.95)
  IDS-SR30 Week 8 | 17.89 (16.19)
Statistical Analysis 1: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < .001, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

13. Other Pre Specified Outcome: High Sensitivity C-Reactive Protein (Hs-CRP)
Description: high sensitivity C-Reactive Protein values will be used to measure inflammation
Time Frame: Baseline and at week 8
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 19
mg/L
  hs-CRP Baseline | 3.56 (8.61)
  hs-CRP Week 8 | 3.72 (9.56)
Statistical Analysis 1: Comparison: Brexpiprazole; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = .295, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Pairwise comparisons were also performed to determine which time points were significantly different from one another

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Brexpiprazole
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 9/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brexpiprazole (N=19)
Restlessness (Nervous system disorders) | 2 (2)
Eye twitch (Eye disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Jaw clenching (Musculoskeletal and connective tissue disorders) | 1 (1)
Weight Gain (Metabolism and nutrition disorders) | 1 (1)
Migraines (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT03427892/Prot_SAP_000.pdf